CLINICAL TRIAL: NCT07291765
Title: Blood Flow Restriction Training in Acute Geriatric Rehabilitation: A Randomized Controlled Trial on Its Effects and Safety in Hospitalized Older Adults.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Principal Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025_A
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia in Elderly

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Blood-Flow-Restriction Training
  Interventions: Device: Stationary Bike + Blood-Flow-Restriction
- Control Group (Active Comparator): Sham-Blood-Flow-Restriction Training
  Interventions: Device: Stationary Bike + Sham-Blood-Flow-Restriction

INTERVENTIONS:
Device: Stationary Bike + Blood-Flow-Restriction — Cycling Intensity individualized + 60% LOP
  Arms: Intervention Group
Device: Stationary Bike + Sham-Blood-Flow-Restriction — Cycling Intensity individualized + 20mmHg
  Arms: Control Group

SUMMARY:
Background: Older adults have a reduced ability to build and maintain muscle mass due to age-related changes in the muscular system. The resulting sarcopenia can lead to a number of health problems and limitations, such as an increased risk of falling and reduced mobility, which can affect quality of life and increase the risk of disease. To increase muscle mass and strength, high-intensity resistance training with loads of 70 to 85% of the repetition maximum (1RM) is recommended. However, this type of training poses a major challenge in the rehabilitation sector, as there is also an increased risk of injury due to physical limitations in old age. According to current research, low-intensity occlusion training could therefore represent a safe and effective training alternative. The aim of this study is therefore to examine the feasibility and effects of blood flow restriction training (BFR) on general health in older adults in a rehabilitative setting.

DETAILED DESCRIPTION:
The study is a randomized controlled trial with a pre-post design. The setting is the premises of St. Marien Hospital in Cologne. Participants will be recruited from the geriatric rehabilitation patient base. Patients will be randomized into 2 groups. The intervention group will be randomly assigned to receive BRF training on an exercise trainer five times a week over a period of two weeks, while the control group will receive sham-BFR training.

ELIGIBILITY:
Inclusion Criteria:

* Adults >65 years with a two week hospitalized acute rehabilitation after a fracture closed to the hip joint

Exclusion Criteria:

* Sickle Cell Anemia
* Iatrogenic changes of the vessels at the place of the tournqiuet application (e.g. Stents)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Pre-Rehabilitation to Post-Rehabilitation (after 2 weeks)
  Isometric Maximal Strength Test of the Knee Extensors (in kg)
Timed Up and Go Test | Pre-Rehabilitation to Post-Rehabilitation (after 2 Weeks)
  The Timed Up and Go Test (TUG) is a widely used English-language assessment for measuring functional mobility and fall risk in older adults. It records the time required to stand up from a chair, walk three meters, turn around, and sit down again.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Marien-Hospital Köln, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No